CLINICAL TRIAL: NCT03554603
Title: Modified Reporting of Positive Urine Cultures Collected From Long Term Care, a Randomized Controlled Trial
Brief Title: Modified Reporting of Positive Urine Cultures Collected From Long Term Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial University of Newfoundland (Other)
Responsible Party: Principal Investigator, Peter Daley, Associate Professor, Memorial University of Newfoundland
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MUN-04
Record Dates: First submitted 2018-06-01; First posted 2018-06-13 (Actual); Results first posted 2024-03-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2023-07

CONDITIONS: Urinary Tract Infections; Asymptomatic Bacteriuria
Keywords: Long term care; Urine culture
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified Reporting (Experimental): Microbiology laboratory will report "Positive urine cultures may represent asymptomatic bacteriuria or urinary tract infection. If urinary tract infection is suspected clinically, please call 777-xxxx (researcher mobile phone) for identification and susceptibility results"
  Interventions: Behavioral: Modified Report
- Standard Reporting (No Intervention): Microbiology laboratory will report identification and susceptibility results

INTERVENTIONS:
Behavioral: Modified Report — An abbreviated version of the microbiology report indicating that growth is present and the physician should call the lab for further details if clinically important.
  Other Names: Restricted Report
  Arms: Modified Reporting

SUMMARY:
Asymptomatic bacteriuria (AB) is a condition in which bacteria are detected in urine culture without urinary symptoms. The inappropriate use of antibiotic treatment for AB selects bacterial flora to express resistance mutations. Reducing inappropriate antibiotic use for AB is difficult, since the microbiology laboratory cannot distinguish patients with AB. The investigators study will use a restricted laboratory report requesting the physician to call the laboratory for culture results. The restricted report may reduce the rate of inappropriate treatment of AB.

DETAILED DESCRIPTION:
Positive urine cultures during the study period will be randomized to restricted microbiology laboratory reporting or standard microbiology laboratory reporting. Physician or patient consent will not be collected. Patient records will be assessed by the investigator to determine if patients have AB or urinary tract infection. Physician antibiotic treatment decision in both groups will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Consecutive positive urine cultures collected from patients admitted to Long term care facilities will be included. All methods of urine collection will be included (midstream, in-and-out catheterization, indwelling catheter).

Exclusion Criteria:

1. Positive urine cultures not collected from Long term care facility patients
2. Pregnancy
3. Antibiotic treatment at the time of collection
4. Patients known to have blood neutrophils <1.0 within 7 days of urine collection

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Health Sciences Center, St. John's, Newfoundland and Labrador, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Modified Reporting | Standard Reporting
Started | 51 | 49
Completed | 49 | 49
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Modified Reporting | Standard Reporting | Total
Number analyzed (Participants) | 51 | 49 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.1 (12.5) | 74.0 (17.7) | 75.0 (15.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 35 | 69
  Male | 17 | 14 | 31
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 51 | 49 | 100
Urinary Tract Infection [Count of Participants; unit: Participants] | 19 | 19 | 38
Asymptomatic Bacteriuria [Count of Participants; unit: Participants] | 32 | 30 | 62

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Asymptomatic Bacteriuria Treated With Antibiotics and Urinary Tract Infection Treated With Antibiotics
Description: Number of Participants Who Received Appropriate Antibiotic Treatment
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Modified Reporting | Standard Reporting
Number analyzed (Participants) | 51 | 49
Participants | 31 | 25

ADVERSE EVENTS:
Time Frame: 30 days
Description: Bacteremia during the trial was considered a serious adverse event
Arm/Group | Modified Reporting | Standard Reporting
All-Cause Mortality (participants affected / at risk) | 2/51 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/51 | 1/49
Other Adverse Events (participants affected / at risk) | 34/51 | 27/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Modified Reporting (N=51) | Standard Reporting (N=49)
Bacteremia (Infections and infestations) | 0 (0) | 1 (1) — Positive blood culture during study period
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Modified Reporting (N=51) | Standard Reporting (N=49)
Tachycardia (Cardiac disorders) | 14 (14) | 8 (8)
Abnormal Temperature (Investigations) | 8 (8) | 5 (5)
Hyperglycemia (Endocrine disorders) | 0 (0) | 1 (1)
Edema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Elevated White Blood Cell Count (Blood and lymphatic system disorders) | 3 (3) | 4 (4)
Altered Mental Status (Nervous system disorders) | 5 (5) | 4 (4)
Tachypnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-01): https://cdn.clinicaltrials.gov/large-docs/03/NCT03554603/Prot_SAP_000.pdf